CLINICAL TRIAL: NCT00585533
Title: A Phase 2 Study of Tarceva for Untreated, Good Prognosis Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI12555; IRB# 00012555; NCT00204724 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other)
  Interventions: Drug: Erlotinib (Tarceva)

INTERVENTIONS:
Drug: Erlotinib (Tarceva) — Erlotinib
  Other Names: Tarceva

SUMMARY:
This study will evaluate Tarceva in a selected population of patients with untreated advanced non-small cell lung cancer who are anticipated to have a relatively good (indolent) prognosis based on clinical criteria. It is anticipated that selection will enrich for tumor characteristic that are likely to be benefited by EGFR inhibitor treatment (survival greater than 90 days). The goal of this strategy is to provide a less toxic, oral treatment for patients with advanced NSCLC that will not interfere with patients receiving chemotherapy at some point in the future and may prolong the time to chemotherapy related progression.

Patients will remain on study until disease progresses, a decline in performance status, if patient cannot tolerate the side effects or develops symptoms requiring conventional chemotherapy.

DETAILED DESCRIPTION:
Primary Objective To determine Time to Chemotherapy Progression (ie includes time on Tarceva monotherapy and chemotherapy) in advanced NSCLC

Secondary Objectives To evaluate survival and response rate associated with Tarceva treatment To study the frequency of symptom improvement (Lung Cancer Subscale)

ELIGIBILITY:
Inclusion Criteria:

* Performance status 0-1.
* Weight Loss < 10% in preceding 3 months
* Age 18 years and older.
* Adjuvant chemotherapy allowed if > 6 months from protocol entry
* Adequate Organ Function
* Liver enzymes < 2X normal, bilirubin = normal
* Oxygen saturation> 89% on room air unless chronically oxygen dependent (not cancer related)
* Creatinine <2.0 mg

Exclusion Criteria:

* Not pregnant or lactating.
* No Clinical Brain Metastases
* No prior chemotherapy for systemic disease
* Imminent need for chemotherapy for impending organ dysfunction is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wallace Akerley, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants enrolled in trial.
Period: Overall Study
Arm/Group | All Participants
Started | 40
Completed | 31
Not Completed | 9
Not completed — objective or symptomatic progression | 9

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (10.09443)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at 6-months Chemotherapy-progression-free (CP-free)
Description: Will determine if 6-month chemotherapy-progression-free (CP-free) survival rate (using RECIST) is significantly higher than the historically observed 31%. A one-sided binomial test at a 5% nominal significance was used.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
percentage of participants | 55 [27.7 to 28.8]

2. Secondary Outcome: Overall Survival
Description: Estimated via a Kaplan-Meier curves. Survival will be counted from the first dose of Tarceva.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | All Participants
Number analyzed (Participants) | 40
weeks | 50.1 [48.5 to 51.7]

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 9/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=40)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Deep Vein Thrombosis (General disorders) | 1 (1)
Paronychia (Skin and subcutaneous tissue disorders) | 2 (2)
Mucositis (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes